CLINICAL TRIAL: NCT06922292
Title: Adaptation, Validity, and Reliability of the Respiratory Distress Observation Scale in Adult Palliative Care Patients: A Turkish Version
Brief Title: "Turkish Validation of the Respiratory Distress Observation Scale in Palliative Care"
Status: Completed | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Elif Kabasakal, LECTURER, Istinye University
Other Study IDs: ISU-2025-001
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-03

CONDITIONS: Dyspnea; Palliative Care; Reliability and Validity
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult Palliative Care Patients With Respiratory Distress: Adult inpatients (≥18 years) receiving palliative care in hospital units, diagnosed with conditions such as lung or pleural cancer, chronic kidney disease, congestive heart failure, COPD, asthma, or pneumonia, and experiencing respiratory distress. Patients must have been staying in the palliative care unit for at least one day and either personally or via a family member provided informed consent to participate in the study.

SUMMARY:
Dyspnea is a subjective experience influenced by physiological, cognitive, behavioral, and sociocultural factors. While self-reported scales are commonly used to assess dyspnea severity, they are unsuitable for patients unable to communicate, such as those with cognitive impairment or sedation. The Respiratory Distress Observation Scale (RDOS), developed by Campbell in 2008, is a reliable and valid tool for evaluating dyspnea in non-communicative palliative care patients. The RDOS has been adapted into Chinese and Italian, but a Turkish version is lacking. This study aims to assess the reliability and validity of the Turkish version of the RDOS.

DETAILED DESCRIPTION:
Any disorder affecting the components of the respiratory system directly impacts respiratory function, while impairments in other systems related to this system indirectly hinder respiratory function. This condition manifests in patients in various ways, including shortness of breath, air hunger, difficulty breathing, a sensation of suffocation, and chest tightness, influenced by physiological, cognitive, behavioral, and sociocultural factors. Under normal conditions, breathing is an unconscious physiological act that goes unnoticed. However, in the presence of the aforementioned disturbances, conscious awareness of the act of breathing emerges. According to the American Thoracic Society (ATS) report, dyspnea is defined as "a subjective experience of breathing discomfort that consists of qualitatively distinct sensations of varying intensity" and is acknowledged as a subjective sensation.

Dyspnea does not result from a single pathophysiological mechanism but may develop due to dysfunctions in multiple systems. Therefore, both identifying the underlying pathophysiology of dyspnea and measuring its presence and severity, given its subjective nature, are of great importance. Dyspnea assessment has been conducted using psychophysical methods and clinical scales. Psychophysical tests measure the perception of respiratory changes in response to externally applied loads, whereas clinical scales aim to determine the magnitude of the work contributing to breathlessness in patients. In addition to identifying the cause of dyspnea and initiating appropriate treatment, accurately measuring dyspnea severity plays a crucial role in planning both medical treatment and pulmonary rehabilitation interventions.

The assessment of dyspnea presence and severity is based on self-reported scales, which are considered partially objective. However, some patients-such as those with cognitive impairment, loss of consciousness, intubation, sedative medication use, or brain injury-are unable to provide self-reports. Monitoring dyspnea in patients unable to self-report has been reported as challenging. In clinical settings, healthcare professionals rely on respiratory rate and oxygen saturation levels to assess dyspnea severity and determine appropriate treatment strategies for such patients.

In Turkey, scales used to assess the presence and severity of dyspnea are based on self-reporting and are therefore not suitable for patients unable to communicate their symptoms. In 2008, Dr. Campbell developed the Respiratory Distress Observation Scale (RDOS) and demonstrated its reliability and validity in patients receiving palliative care-such as those with cancer, chronic obstructive pulmonary disease (COPD), heart failure, and pneumonia-who are unable to self-report their dyspnea. The RDOS consists of eight indicators related to dyspnea and takes less than five minutes to administer. Originally developed in English, the RDOS has been translated into Chinese and Italian. However, a Turkish version of the scale is needed. This study aims to examine the reliability and validity of the Turkish version of the RDOS.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older,
* Diagnosed with lung or pleural cancer, chronic kidney failure, congestive heart failure, COPD, asthma, or pneumonia, and experiencing dyspnea,
* Specifically referred for treatment of dyspnea,
* Residing in a palliative care unit for at least 1 day,
* Willing to participate in the study, either personally or through consent from a family member.

Exclusion Criteria:

* Completely dependent on a ventilator,
* Diagnosed with a central nervous system disorder (Quadriplegia, Bulbar ALS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving inpatient treatment in the Intensive Care Unit who meet the inclusion criteria will be included in the study. The relatives of eligible patients will be informed about the study, and informed consent will be obtained. The study will be conducted in accordance with the principles of the Helsinki Declaration and Good Clinical Practice guidelines. Participants included in the study will be assigned a unique code (based on date of birth and order of participation).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Respiratory Distress Observation Scale (RDOS) | Within the first assessment (Day 1) and repeated measures within 2 hours after baseline assessment
  The RDOS was developed by Campbell to measure the presence and intensity of respiratory distress for patients who are unable to self-report dyspnea. The eight parameters assessed by the observer are assess heart rate, respiratory, restlessness, paradoxical breathing pattern, accessory muscle use, grunting at end-expiration, nasal flaring, and look of fear. Four parameters scored between 0 and 2 points; the other four parameters scored 0, or 2 points and progressed from most to least severity of distress. The intensity of respiratory distress is reflected by a total score ranging from 0 to 18. A high total score increases the risk of developing respiratory distress. RDOS score of 0 to 2 suggests no respiratory distress; a score of 3, mild distress; scores of 4 to 6, moderate distress; and 7 or greater, severe distress, with an adequate cutoff point for assigning clinical significance at a score of 3.

SECONDARY OUTCOMES:
Heart Rate Assessment | Within 30 minutes prior to RDOS administration
  Heart rate (beats per minute) will be extracted from patient records within 30 minutes before the RDOS (Respiratory Distress Observation Scale) assessment.
Systolic Blood Pressure Assessment | Within 30 minutes prior to RDOS administration
  Systolic blood pressure (mmHg) will be recorded from clinical documentation within 30 minutes before RDOS administration.
Diastolic Blood Pressure Assessment | Within 30 minutes prior to RDOS administration
  Diastolic blood pressure (mmHg) will be obtained from the patient's chart and used as a physiological indicator at the time of RDOS evaluatio
Respiratory Rate Assessment | Within 30 minutes prior to RDOS administration
  Respiratory rate (breaths per minute) will be noted from medical records as a clinical vital sign prior to RDOS assessment.
Oxygen Saturation Assessment | Within 30 minutes prior to RDOS administration
  Peripheral oxygen saturation (SpO₂, %) will be documented from the monitoring system or medical record shortly before RDOS scoring.
Body Temperature Assessment | Within 30 minutes prior to RDOS administration
  Body temperature (°C) will be recorded from the most recent measurement available before the RDOS is administered.
Partial Pressure of Oxygen (PaO₂) Assessment | Within 30 minutes prior to RDOS administration
  The most recent arterial partial pressure of oxygen (PaO₂, mmHg) will be obtained from medical records. The sample must be collected within 30 minutes prior to RDOS assessment.
Partial Pressure of Carbon Dioxide (PaCO₂) Assessment | Within 30 minutes prior to RDOS administration
  Arterial partial pressure of carbon dioxide (PaCO₂, mmHg) will be recorded from laboratory results. The value must be based on a sample taken no more than 30 minutes before RDOS administration.
Arterial Oxygen Saturation (SaO₂) Assessment | Within 30 minutes prior to RDOS administration
  SaO₂ (%) will be documented from arterial blood gas analysis and used as an objective indicator of blood oxygenation status.
Blood pH Assessment | Within 30 minutes prior to RDOS administration
  Arterial blood pH values will be extracted from the most recent arterial blood gas test, conducted within 30 minutes prior to RDOS application.
Bicarbonate (HCO₃-) Assessment | Within 30 minutes prior to RDOS administration
  The bicarbonate (HCO₃-, mmol/L) level will be obtained from arterial blood gas test results and analyzed as part of metabolic status assessment.
Dyspnea Assessment | At baseline
  Verbal Dyspnea Scale (VDS):Conscious patients will self-rate their level of breathlessness on a 0-10 numeric rating scale, where 0 indicates no dyspnea and 10 indicates the most severe dyspnea.
ICU Stay Duration | At enrollment
  Duration of stay in the intensive care unit (ICU) will be recorded in days from hospital records.
Glasgow Coma Scale (GCS) Assessment | At enrollment
  The Glasgow Coma Scale score will be recorded to assess the participant's level of consciousness. The Glasgow Coma Scale (GCS) will be used to determine the patient's level of consciousness. The Glasgow Coma Scale (GCS) assesses consciousness by evaluating three components: eye opening (4-1), verbal response (5-1), and motor response (6-1). Scores range from 3 (deep coma) to 15 (fully alert), with lower scores indicating more severe impairment. A score of 8 or below typically suggests the need for immediate intervention.
Clock Drawing Test Assessment | At enrollment
  Cognitive function will be assessed using the Clock Drawing Test, scored based on spatial and time-setting accuracy.
Palliative Performance Scale (PPS) Score Assessment | At enrollment
  The Palliative Performance Scale (PPS) is a validated clinical tool used to assess the functional status of patients receiving palliative care. It ranges from 0% (death) to 100% (fully active) in 10% increments, based on five parameters: ambulation, activity level and extent of disease, self-care ability, oral intake, and level of consciousness. A high PPS score (e.g., 80-100%) indicates that the patient is active, independent, and has minimal care needs, while a low PPS score (e.g., 10-30%) reflects a patient who is bedbound, has limited intake and consciousness, and requires full care. PPS is widely used to estimate survival time, guide care planning, and classify patients in clinical research. Lower scores are associated with reduced life expectancy and higher dependency.
Type of Respiratory Support Assessment | At enrollment
  The type of respiratory support (e.g., High-Flow Oxygen [HFO], Non-Invasive Mechanical Ventilation [NIMV], Invasive Mechanical Ventilation [IMV]) used at the time of RDOS assessment will be documented.
Fraction of Inspired Oxygen (FiO₂) Assessment | At baseline
  FiO₂ (%) values will be documented from respiratory support devices to assess oxygen delivery.
PaO₂/FiO₂ Ratio Assessment | At baseline
  The ratio of arterial oxygen pressure (PaO₂) to inspired oxygen fraction (FiO₂) will be calculated to assess oxygenation efficiency.

CONTACTS AND LOCATIONS:
Locations (1):
- Istınye University, Istanbul,, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Tinti S, Destrebecq A, Terzoni S, De Maria B, Falcone G, Da Col D, Pairona G, Longhi C, Giudici E, Pidone IM, Alberti A, Sofia M, Ramponi I, Campbell ML. Respiratory Distress Observation Scale Italian Version: Cultural-Linguistic Validation and Psychometric Properties. J Hosp Palliat Nurs. 2021 Apr 1;23(2):187-194. doi: 10.1097/NJH.0000000000000736. PMID 33633100
- [Background] Pianosi PT, Zhang Z, Hernandez P, Huebner M. Measuring Dyspnea and Perceived Exertion in Healthy Adults and with Respiratory Disease: New Pictorial Scales. Sports Med Open. 2016;2:17. doi: 10.1186/s40798-015-0038-4. Epub 2016 Jan 7. PMID 26770885
- [Background] Eakin EG, Resnikoff PM, Prewitt LM, Ries AL, Kaplan RM. Validation of a new dyspnea measure: the UCSD Shortness of Breath Questionnaire. University of California, San Diego. Chest. 1998 Mar;113(3):619-24. doi: 10.1378/chest.113.3.619. PMID 9515834
- [Background] Parshall MB, Schwartzstein RM, Adams L, Banzett RB, Manning HL, Bourbeau J, Calverley PM, Gift AG, Harver A, Lareau SC, Mahler DA, Meek PM, O'Donnell DE; American Thoracic Society Committee on Dyspnea. An official American Thoracic Society statement: update on the mechanisms, assessment, and management of dyspnea. Am J Respir Crit Care Med. 2012 Feb 15;185(4):435-52. doi: 10.1164/rccm.201111-2042ST. PMID 22336677
- [Result] Ambrosino N, Porta R. Measurement of dyspnoea. Monaldi Arch Chest Dis. 2001 Feb;56(1):39-42. PMID 11407208
- [Result] Dyspnea. Mechanisms, assessment, and management: a consensus statement. American Thoracic Society. Am J Respir Crit Care Med. 1999 Jan;159(1):321-40. doi: 10.1164/ajrccm.159.1.ats898. No abstract available. PMID 9872857
- [Result] Coccia CB, Palkowski GH, Schweitzer B, Motsohi T, Ntusi NA. Dyspnoea: Pathophysiology and a clinical approach. S Afr Med J. 2016 Jan;106(1):32-6. doi: 10.7196/samj.2016.v106i1.10324. PMID 26933707